CLINICAL TRIAL: NCT07148258
Title: Evaluating Georgia Part C Implementation Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Georgia Department of Public Health (Unknown)
Responsible Party: Principal Investigator, Katherine E. Pickard, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00010098; 1K23MH130651-01A1 (NIH); 2025P013101 (Other: Emory IRB)
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Communication Disorder, Childhood; Autism
Keywords: Caregivers; Early Intervention (EI) Providers; Early Intervention System; Project ImPACT; Social communication delays
MeSH Terms: conditions — Communication Disorders; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Intervention (EI) providers (Other): Early Intervention (EI) providers who serve young children with social communication delays and/or autism will report on their experiences delivering Project ImPACT via one of two training models. Providers will have the option of consenting to share videos of their Project ImPACT sessions to help us understand the quality of Project ImPACT delivery.
  Interventions: Other: Project ImPACT Training As Usual; Other: Project ImPACT Training Plus Co-Production
- Caregivers (Other): Caregivers of children under 36 months of age in the Georgia EI system who are receiving services within the EI system will report on their experiences with the providers who have been trained in one of the two Project ImPACT models.
  Caregivers will either: 1) complete surveys before and after they receive Project ImPACT, or 2) complete a confidential survey after receiving Project ImPACT from their provider. Caregivers will have the option of consenting to share videos of their Project ImPACT sessions to help us understand the quality of Project ImPACT delivery.
  Interventions: Behavioral: Routine Project ImPACT

INTERVENTIONS:
Other: Project ImPACT Training As Usual — Project ImPACT is an evidence-based autism intervention that teaches parents to use a blend of developmental and naturalistic behavioral intervention techniques across a variety of daily routines to enhance their child's social engagement, language, imitation, and play skills.
  The typical training model for Project ImPACT includes a 6-hour, interactive online tutorial that walks providers through the core Project ImPACT intervention strategies. After completing the online tutorial, providers attend a live interactive workshop virtually that is spread across 4, 3.5-hour days (14 hours total). Providers receive 1 hour of consultation once every other week for an hour from a trained Project ImPACT consultant (research staff member) following training.
  Other Names: Usual ImPACT
  Arms: Early Intervention (EI) providers
Other: Project ImPACT Training Plus Co-Production — Project ImPACT is an evidence-based autism intervention that teaches parents to use a blend of developmental and naturalistic behavioral intervention techniques across a variety of daily routines to enhance their child's social engagement, language, imitation, and play skills.
  The second cohort for Project ImPACT training is a model in which providers receive the same typical Project ImPACT training activities, in addition to three supplemental modules on other common areas of concern for families and how best to integrate other topics within Project ImPACT to meet the diverse needs of families.
  Other Names: Usual ImPACT + Supplements
  Arms: Early Intervention (EI) providers
Behavioral: Routine Project ImPACT — Project ImPACT is an evidence-based autism intervention that teaches parents to use a blend of developmental and naturalistic behavioral intervention techniques across a variety of daily routines to enhance their child's social engagement, language, imitation, and play skills. Project ImPACT is delivered with parents meeting once or twice each week for one hour over 12- 16 weeks. In each session, parents receive: 1) didactic instruction in intervention strategies; 2) modeling of the intervention techniques by the therapist; 3) live coaching from the therapist while practicing the strategies with their child; and 4) homework to practice the strategies at home with their child, 20 minutes each day across meaningful home routines.
  Arms: Caregivers

SUMMARY:
This study aims to answer the question: What is the best way to help Early Intervention (EI) providers deliver high-quality services to children with communication delays for autism?

The primary goal of this project is to examine the outcomes associated with delivering Project ImPACT, an evidence-based autism intervention that is delivered as part of routine training within Georgia's EI system. Providers in the study will receive one of two Project ImPACT training models to help us understand which training model helps providers learn Project ImPACT better. Specifically, this study will examine the: 1) the process and quality by which Project ImPACT is implemented and adapted by EI providers across the two training conditions; 2) factors that impact how well Project ImPACT is implemented; and 3) the child (i.e., social communication) and family (i.e., parent empowerment and fidelity) outcomes associated with receiving Project ImPACT.

DETAILED DESCRIPTION:
This study aims to determine the: 1) implementation outcomes; and 2) preliminary parent and child outcomes associated with Project ImPACT when implemented within the Georgia Early Intervention (EI) system. 150 EI providers will be trained in one of two Project ImPACT training models. Training will include the option for group consultation. This training is part of standard training requirements, so it is not considered research.

Participating caregivers who receive Project ImPACT will receive the program as part of their routine EI services. They will have two options to participate in this research: 1) complete surveys before and after participation in Project ImPACT (each set will take 20-30 minutes), as well as an exit interview; or 2) complete a confidential survey only after participating in Project ImPACT, which will take 20-30 minutes. All research activities will be conducted at the Marcus Autism Center.

ELIGIBILITY:
Inclusion Criteria for Providers:

* Currently employed or contracted by Georgia's EI system
* Maintain an active therapy caseload
* Fluent in English.

Inclusion Criteria for Caregivers:

* Have a child under 36 months currently enrolled in services through Georgia's Early Intervention system
* Are being seen by a provider participating in Project ImPACT training and research
* Fluent in English.

Exclusion Criteria for both Providers and Caregivers:

* Not meeting the eligibility criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Project ImPACT Coaching Fidelity | Biweekly up to 20 weeks
  Providers' Project ImPACT therapy sessions will be video recorded and will be scored retrospectively for use of core Project ImPACT strategies. The research team will measure the project fidelity by watching recorded videos of the sessions, which will allow the team to capture how effectively the adult implements a strategy. This will be scored using the Project ImPACT fidelity checklist. Provider fidelity for each intervention strategy will be rated by a trained coder using a 5-point Likert scale, with scores of 4 or greater indicating appropriate fidelity. An average score of 4 or higher on all of the strategies indicates that fidelity has been met for Project ImPACT.
Provider Co-Production Quality | Baseline; Weekly up to 12 weeks, and 6-months
  Following each therapy session, providers will complete a brief 20-item survey in which they will be asked what their session looked like and the rationale for any adaptations described. Providers will first indicate how long in minutes their Project ImPACT session was. They will also indicate which Project ImPACT coaching activities they completed in their session (yes/no). Providers will then be asked to indicate which of 10 additional non-Project ImPACT topics they covered in their session and subsequently how long in minutes they spent covering the additional topics. The following information will then be calculated for each session: 1) Percent of possible coaching elements delivered; 2) Percent of time spent covering additional topics; 3) Percent of time delivering other topics.

SECONDARY OUTCOMES:
Project ImPACT Self-Efficacy. | Baseline, 1-month after baseline (post-Project ImPACT training), and 12 months
  Providers will rate their self-efficacy using a 7-item measure that asks about their perceived skills delivering Project ImPACT core strategies. Providers will rate each item using a 10-point Likert scale (1 = not at all confident, 5 = somewhat confident, and 10 = completely confident). An increase in the mean score indicates that the intervention has successfully enhanced self-efficacy.
Perceived Characteristics of the Intervention Scale (Project ImPACT Perceptions) | Study completion (on average 12 months)
  All providers will complete the Perceived Characteristics of the Intervention Scale (PCIS). The PCIS is a 12-item questionnaire that measures the perceived characteristics of an intervention that are thought to impact its uptake and use. The current study will use an abbreviated measure that includes the following dimensions: Relative Advantage (e.g., "Project ImPACT is more effective than other therapies I have used"), Compatibility (e.g., "Project ImPACT is aligned with my clinical judgement"), Complexity (e.g., "Project ImPACT is easy to use"), and Potential for Reinvention (e.g., "Project ImPACT can be adapted to meet the needs of my patients"). Participants will rate each item on a 7-point Likert scale (1 = Strongly disagree, 7 = Strongly agree). Higher scores generally indicate more positive perceptions of the intervention.
The Family Outcome Survey (caregivers) | Baseline and study completion (on average 6 months)
  The Family Outcome Survey (FOS) measures family outcomes expected to change through participation in early intervention programs for children with disabilities and their caregivers. The FOS includes five outcomes: understanding your child's strengths, needs, and abilities; knowing your rights and advocating for your child; helping your child develop and learn; having support systems; and accessing the community. The FOS comprises 24 items, with four to six items per outcome. Responses range from not at all (1) to completely (5). To get overall scores, all the responses are summed for the items within each of the five outcome areas and the three helpfulness indicators.
  The Early Childhood Technical Assistance (ECTA) Center recommends that scores of 5 or greater on the family outcome items be considered an indicator of outcome attainment. Scores below 5 may indicate areas requiring further improvement
Parent Observation of Social Interaction | Baseline
  Parent Observation of Social Interaction (POSI). The POSI is a 7-item measure that asks caregivers to rate their child's use of social communication skills, including communication, gesturing, and play, with each question scored as either 0 or 1. A score of 3 or more indicates a positive screen, suggesting the child may be at risk and warrants further evaluation.
Social Communication Checklist (caregivers) | Baseline and study completion (on average 6 months)
  Social Communication Checklist (SCC). The SCC was developed as part of the Project ImPACT curriculum. The SCC is a 70-item checklist; respondents indicate if a child uses each skill, "Rarely/Not Yet (1)," "Sometimes, but not consistently (2)," or "Usually, at least 75% of the time (3)." Items correspond with the social communication domains targeted in Project ImPACT: 10 social engagement items, 24 language/ communication items, and 13 imitation/play items, and were summed for domain scores and a Total Score. Each item reflecting abnormal behavior scores 1 point; others score 0.
  Total Scores: Range from 0 to 39 for verbal children and 0-33 for nonverbal children. Higher scores indicate greater social communication impairment.
Project ImPACT Fidelity for Parents. | Baseline and study completion (on average 6 months)
  The project fidelity for Parent behavior will be scored for correct use of the Project ImPACT intervention techniques during the first and final Project ImPACT sessions using the Project ImPACT fidelity checklist. Parent fidelity for each intervention strategy will be rated by a trained coder using a 5-point Likert scale, with scores of 4 or greater indicating appropriate fidelity.
Project ImPACT Satisfaction. | Study completion (on average 6 months)
  All parents will complete a 16-item survey examining: 1) treatment acceptability; 2) perceived child social communication gains; 3) burden of the treatment on the family; and 4) frequency of program use. Parents will rate their agreement with statements reflecting these domains on a 7-point Likert scale (ranging from "Completely dissatisfied" to "Completely satisfied," with a neutral midpoint and intermediate options in between). A higher score indicates a higher level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E. Pickard, PhD, Principal Investigator — Emory University
Locations (1):
- Marcus Autism Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share the data related to the primary study outcomes and study protocol.
Supporting Information: Study Protocol
Time Frame: Data will be shared by the research team after the study has been completed.
Access Criteria: The research team will share the data through the NIH's NDAR (National Database for Autism Research).